CLINICAL TRIAL: NCT04104425
Title: Role of Lactate Level in Prediction of Patients'Acute Gastrointestinal Bleeding Admissions to Intensive Care Unit, Interventions and Short Term Outcomes
Brief Title: Lactate Level and Gastrointestinal Bleeding
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hekmat Nashat Shawky Zakhary, principal invistigator, Assiut University
Other Study IDs: LA in GIB
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Patient Compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute gastrointestinal bleeding is a common emergency with significant morbidity, mortality, and cost. Appropriate risk stratification of patients presenting with acute gastrointestinal bleeding aids in the triage of patients to determine need for hospital admission and the need for emergency endoscopic intervention. Increased blood lactate levels are common in critically ill patients. Our study will evaluate the usefulness of lactate measurements on resources utilisation ( intensive care unit admission, length of hospital stay) and other patient-oriented outcomes ( need for transfusion and endoscopy) in patients with acute gastrointestinal bleeding.

DETAILED DESCRIPTION:
The present study is a prospective cross sectional study aimed to assess whether venous blood lactate on hospital presentation is predictive of need for interventions and short term outcomes (eg PRBC transfusion, ICU admission ) in patients with acute GIB who presented to ED of Assuit University hospital between September 2019 and June 2022. The study included 300 patients with acute GIB. Out of those patients; 200 patients had elevated blood lactate and 100 patients had normal blood lactate.

It was found that mean age of patients with elevated lactate was significantly higher in comparison to those with normal lactate. There were no significant differences between both groups as regard risk factors for bleeding (use of anti-coagulants, aspirin), use of NSAIDs was higher among patients with normal lactate while history of prior UGIB was higher among patients with elevated lactate. The most frequent presentations among the studied patients were hematemesis and melena.

Both groups had insignificant differences as regard laboratory data, endoscopic findings and interventions.

Patients with elevated lactate had prolonged hospital stay, higher frequency of blood transfusion, ICU admission and mortality in comparison to those with normal blood lactate.

Based on the current study, predictors of mortality among patients with UGIB were old age , LC, elevated lactate and variceal bleeding.

So we could say that elevated blood lactate can be predictive for interventions and short term outcomes in patients with acute GIB ,however, further and similar studies with multi-center settings would be more reliable and accurate.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with acute gastrointestinal bleeding, inclusive of both upper and lower sources
* Patients ≥18 years old

Exclusion Criteria:

* Patients with tumor bleeding
* patients with post procedure or surgical site bleeding
* patients with active systemic infection
* patients wit post-cardiopulmonary resuscitation state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with acute gastrointestinal bleeding to emergency department of Assiut University hospital
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
The need for intensive care unit admissions, intervention and short term outcomes ( packed red blood cells transfusion) in patients with acute gastrointestinal bleeding and elevated lactate level | 2 years
  Assessment of role of elevated lactate level in predicting the need for intensive care unit admissions, emergency endoscopic intervention and packed red blood cells transfusion in patients with acute gastrointestinal bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Result] Zippi M, Febbraro I, De Felici I, Mattei E, Traversa G, Occhigrossi G. [Diagnosis and treatment of bleeding peptic ulcer: our experience]. Clin Ter. 2008 Jul-Aug;159(4):249-55. Italian. PMID 18776982
- [Result] Musikatavorn K, Thepnimitra S, Komindr A, Puttaphaisan P, Rojanasarntikul D. Venous lactate in predicting the need for intensive care unit and mortality among nonelderly sepsis patients with stable hemodynamic. Am J Emerg Med. 2015 Jul;33(7):925-30. doi: 10.1016/j.ajem.2015.04.010. Epub 2015 Apr 10. PMID 25936479
- [Result] Shah A, Chisolm-Straker M, Alexander A, Rattu M, Dikdan S, Manini AF. Prognostic use of lactate to predict inpatient mortality in acute gastrointestinal hemorrhage. Am J Emerg Med. 2014 Jul;32(7):752-5. doi: 10.1016/j.ajem.2014.02.010. Epub 2014 Feb 17. PMID 24813902
- [Result] El-Kersh K, Chaddha U, Sinha RS, Saad M, Guardiola J, Cavallazzi R. Predictive Role of Admission Lactate Level in Critically Ill Patients with Acute Upper Gastrointestinal Bleeding. J Emerg Med. 2015 Sep;49(3):318-25. doi: 10.1016/j.jemermed.2015.04.008. Epub 2015 Jun 22. PMID 26113379
- [Result] Wada T, Hagiwara A, Uemura T, Yahagi N, Kimura A. Early lactate clearance for predicting active bleeding in critically ill patients with acute upper gastrointestinal bleeding: a retrospective study. Intern Emerg Med. 2016 Aug;11(5):737-43. doi: 10.1007/s11739-016-1392-z. Epub 2016 Feb 2. PMID 26837207
- [Result] Shrestha MP, Borgstrom M, Trowers EA. Elevated lactate level predicts intensive care unit admissions, endoscopies and transfusions in patients with acute gastrointestinal bleeding. Clin Exp Gastroenterol. 2018 May 23;11:185-192. doi: 10.2147/CEG.S162703. eCollection 2018. PMID 29872331
- [Result] Hernandez G, Bruhn A, Castro R, Regueira T. The holistic view on perfusion monitoring in septic shock. Curr Opin Crit Care. 2012 Jun;18(3):280-6. doi: 10.1097/MCC.0b013e3283532c08. PMID 22473257